CLINICAL TRIAL: NCT02172872
Title: 10-day Decitabine Versus Conventional Chemotherapy ("3+7") Followed by Allografting in AML Patients ≥ 60 Years: a Randomized Phase III Study of the EORTC Leukemia Group, CELG, GIMEMA and German MDS Study Group
Brief Title: "InDACtion" vs "3+7" Induction in AML
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Janssen Pharmaceuticals (Industry); Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-1301; 2014-001486-27 (EudraCT Number)
Record Dates: First submitted 2014-06-19; First posted 2014-06-24 (Estimated); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Acute Myeloid Leukemia (AML)
Keywords: Newly diagnosed; AML; Elderly; Decitabine; Transplant
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- standard combination chemotherapy (Active Comparator)
  Interventions: Drug: standard combination chemotherapy
- decitabine (Experimental)
  Interventions: Drug: decitabine

INTERVENTIONS:
Drug: standard combination chemotherapy — 1. Cycle 1
     1. daunorubicin (60 mg/m²) infusion (15-30 min) for 3 days
     2. cytarabine (200 mg/m²) continuous infusion (24 hrs) for 7 days.
  2. Cycle 2
     1. daunorubicin (45 mg/m²) infusion (15-30 min) for 3 days
     2. cytarabine (200 mg/m²) continuous infusion (24 hrs) for 7 days.
  3. Cycle 3 (mini-ICE)
     1. idarubicin (8 mg/m²) infusion (15-30 min) for 3 days
     2. cytarabine (100 mg/m²) continuous infusion (24 hrs) for 5 days
     3. etoposide (100 mg/m²) infusion (1 hr) for 3 days
  4. Cycle 4 (mini-ICE) (optional)
     1. idarubicin (8 mg/m²) infusion (15-30 min) for 3 days
     2. cytarabine (100 mg/m²) continuous infusion (24 hrs) for 5 days
     3. etoposide (100 mg/m²) infusion (1 hr) for 3 days
  Other Names: "3+7" induction chemotherapy; Intensive combined chemotherapy
  Arms: standard combination chemotherapy
Drug: decitabine — 1. Cycle 1: decitabine (20 mg/m²) infusion (1 hr) for 10 days
  2. Cycle 2
     1. if bone marrow (BM) blasts < 5%: decitabine (20 mg/m²) infusion (1 hr) for 5 days
     2. if BM blasts >= 5%: decitabine (20 mg/m²) infusion (1 hr) for 10 days
  3. Cycle 3
     1. if BM blasts < 5%: decitabine (20 mg/m²) infusion (1 hr) for 5 days
     2. if BM blasts >= 5%: decitabine (20 mg/m²) infusion (1 hr) for 10 days
  4. Cycle 4-6: decitabine (20 mg/m²) infusion (1 hr) for 5 days
  5. Continuation therapy from Cycle 7 and until 'progression or toxicity': decitabine (20 mg/m²) infusion (1 hr) for 5 days or 3 days
  Note: All patients considered eligible for transplant should be consolidated with alloHCT once donor is available.
  Other Names: Dacogen
  Arms: decitabine

SUMMARY:
Older patients with acute myeloid leukemia (AML) have a small (< 10%) chance of long-term survival. Despite the treatment of elderly AML patients with intensive chemotherapy, the survival has not been improved during the last decades.

The purpose of this study is to determine whether frontline therapy with a 10-day decitabine schedule provides a better survival than standard intensive combination chemotherapy in elderly AML patients (>= 60 years).

DETAILED DESCRIPTION:
* The overall survival (OS) of older AML patients has not been improved during the last decades with intensive chemotherapy based on cytarabine combined with an anthracycline ("3+7").
* Next generation sequencing technology reveals that mutations in genes involved in epigenetics are frequently mutated in AML (e.g. DNMT3a), suggesting an important role of epigenetics in the pathophysiology of AML. Decitabine (given in a 5-day schedule) has been shown to be superior to low-dose Ara-C.
* A retrospective analysis revealed that epigenetic therapy (either azacitidine or decitabine) is associated with similar survival rates as intensive chemotherapy in older patients (n=671) with newly diagnosed AML.
* The recently published encouraging phase 2 data with the 10-day decitabine schedule suggests that decitabine results in similar CR rates compared with intensive chemotherapy. Allogeneic transplantation (alloHCT) also offers the opportunity for cure among older AML patients, therefore treatment strategies should aim to allograft older AML patients.
* Decitabine treatment can lead to very interesting cure rates when used as "bridging" to allografting.

Based on the data summarized above, we hypothesize that decitabine at a daily dose of 20 mg/m² starting with the 10-day schedule followed by an alloHCT or by continuation of 5-days decitabine cycles is superior to conventional intensive chemotherapy in older AML patients.

ELIGIBILITY:
Inclusion criteria:

1. Age ≥ 60 years
2. WHO Performance status ≤ 2
3. Eligible for standard intensive chemotherapy
4. Newly diagnosed AML cytopathologically confirmed to the WHO classification (up to 2 months prior to randomization)
5. De novo or secondary AML is allowed
6. White blood cell (WBC) count is ≤ 30x10E9/L (measured within 72 hours prior to randomization).
7. Laboratory assessments (measured prior to randomization):

   1. serum glutamate oxaloacetate transaminase (SGOT / ASAT) and serum glutamate pyruvate transaminase (SGPT / ALAT) < 2.5 x the upper limit of normal range unless considered AML-related
   2. Total serum bilirubin < 2.5 x the upper limit of normal range unless considered AML-related or due to Gilbert's syndrome
   3. Serum creatinine < 2.5 x the upper limit of normal range unless considered AML-related
8. Patients of reproductive potential should use adequate birth control measures, as defined by investigator, during the study treatment period and for at least 3 months after the last study treatment.
9. Before patient registration/randomization, written informed consent must be given according to the International Conference of Harmonization good clinical practice (ICH GCP) and national/local regulations

Exclusion criteria:

1. Presence of acute promyelocytic leukemia (APL, i.e. AML-M3 with t(15;17)(q22;q12); promyelocytic leukemia - retinoic acid receptor-alpha (PML-RARA) fusion gene and cytogenetic variants)
2. Presence of blast crisis of chronic myeloid leukemia
3. Presence of active central nervous system (CNS) leukemia
4. Patients did not receive any prior treatment for AML (relapsed AML is not allowed), such as any antileukemic therapy including investigational agents and hypomethylating agents (decitabine, 5-azacytidine). Treatment with hydroxyurea (HU) is allowed to control the leukocytosis if given preferably for less than 5 days and is stopped at least two days prior to the start of any of the protocol regimens
5. Patients received any prior treatment for myelodysplastic syndrome (MDS) or myeloproliferative neoplasms (MPN) with:

   1. hypomethylating agents (decitabine, 5-azacytidine), OR
   2. with intensive chemotherapy or transplantation within the last three years
   3. NOTE: The following treatments for previous MDS or MPN are allowed (up to one month before inclusion):

      * Growth factors, thrombomimetics, immunosuppression (cyclosporin A, steroids, antithymocyte globulin etc.), chelation, interferons, anagrelide
      * Lenalidomide, low-dose chemotherapy (low-dose melphalan, HU, low-dose cytarabine etc.), tyrosine-kinase inhibitors, histone deacetylase inhibitors (e.g. valproic acid, panobinostat etc.), mammalian target of rapamycin (mTOR) inhibitors, other experimental treatment that is not based on inhibition of deoxyribonucleic acid (DNA) methyltransferase
6. Presence of concomitant severe cardiovascular disease which would make intensive chemotherapy impossible, i.e. uncontrolled arrhythmias requiring chronic treatment, congestive heart failure or symptomatic ischemic heart disease, reduced left ventricular function assessed by multigated acquisition (MUGA) scan or echocardiogram
7. Presence of any malignancy (except basal and squamous cell carcinoma of the skin) for which the patient received systemic anticancer treatment within 6 months prior to randomization NOTE: Diagnosis of any previous or concomitant malignancy is thus not an exclusion criterion.
8. Presence of active uncontrolled infection
9. Presence of any psychological, familial, sociological or geographical condition in the opinion of the investigator potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 606 (Actual)
Dates: Start 2014-11-28 (Actual); Primary Completion 2022-03-07 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | 4.9 years from first patient in

SECONDARY OUTCOMES:
Occurrence of adverse events (AEs) | 4.9 years from first patient in
  The events are graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0
Progression-free survival (PFS) from randomization to the date of either first progression, first relapse or death, whichever occurs first | 4.9 years from first patient in
Transplantation feasibility | 4.9 years from first patient in
  Percentage of patients transplanted
Outcome post-transplantation | 4.9 years from first patient in
  PFS, incidence of relapse or progression, and incidence of non-relapse or progression related mortality
Health economics impact of each treatment arm | 4.9 years from first patient in
  At the end of each cycle, duration of hospitalization and number of visits (planned or related to event), number of transfusions, growth factor support and intravenous anti-infective are collected
Health Related Quality of Life (HRQoL) questionnaires | 4.9 years from first patient in
  EORTC Quality of Life Questionnaire (QLQ-C30) Elderly module (ELD14)
Prognostic value of baseline physical and functional conditions on treatment outcome using geriatric assessment tools | 4.9 years from first patient in
  Short physical performance battery (SPPB) and activities of daily living (ADL)
complete response (CR/CRi) rate | 4.9 years from first patient in
  All patients who reached complete response (CR) or complete response with incomplete marrow recovery (CRi) after the administration of protocol treatment ("3+7" or decitabine)
Overall CR/CRi rate | 4.9 years from first patient in
  All patients who reached CR or CRi, after administration of the protocol treatment ("3+7" or decitabine) or following another salvage/new treatment for AML (other than transplant)
Disease-free survival (DFS) from CR or CRi | 4.9 years from first patient in
  The time between the date of CR or CRi and the date of first relapse or death (whatever the cause), whichever occurs first

CONTACTS AND LOCATIONS:
Overall Officials: Michael Luebbert, MD, PhD, Study Chair — Universitaetsklinikum Freiburg, Freiburg, Germany; Gerwin G Huls, MD, PhD, Principal Investigator — UMCG, Groningen, The Netherlands; Pierre W Wijermans, MD, Principal Investigator — HagaZiekenhuis, the Hague, The Netherlands
Locations (53):
- Belgium (7):
  - UZ Antwerpen, Edegem, Antwerpen
  - UZ Brussel, Jette, Brussels Capital
  - CHR Verviers, Verviers, Liège
  - A.Z. St. Jan, Bruges, West-Vlaanderen
  - Institut Jules Bordet, Brussels
  - C.H.U. Sart-Tilman, Liège
  - CHR De La Citadelle, Liège
- National Specialized Hospital for Active Treatment of Haematological Diseases, Sofia, Bulgaria
- Croatia (2):
  - Clinical Hospital Merkur, Zagreb
  - University Hospital Rebro, Zagreb
- France (3):
  - CHU de Caen - Hôpital Côte de Nacre, Caen
  - CHU de Nantes - Hôtel Dieu, Nantes
  - Assistance Publique - Hôpitaux de Paris - Hôpital Saint Antoine, Paris
- Germany (9):
  - Universitätsklinikum Aachen AÖR - Medizinische Fakultät der RWTH, Aachen
  - Klinikum Augsburg, Augsburg
  - Helios Kliniken - Helios Klinikum Berlin-Buch, Berlin
  - Universitätsklinikum Essen, Essen
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Universitaetklinikum Halle - Martin Luther Universitaet - Universitaetsklinikum Halle (Saale), Halle
  - Klinikum Der Phillips - Universität Marburg, Marburg
  - Universitaet Rostock - Medizinische Fakultaet, Rostock
  - Universitaetsklinikum Tuebingen-Uni Kliniken Berg, Tübingen
- Italy (21):
  - Azienda Ospedaliero Universitaria - Ospedali Riuniti, Ancona
  - Universita Degli Studi Di Bari - Policlinico, Bari
  - Universita di Bologna, Bologna
  - Ospedale Regionale A. Pugliese, Catanzaro
  - Ospedali Riuniti Foggia, Foggia
  - Azienda Ospedaliero - Universitaria Policlinico di Modena, Modena
  - Amedeo Avogadro University of Eastern Piedmont-Ospedale Maggiore della Carita, Novara
  - La Maddalena S.P.A., Palermo
  - Ospedale San Salvatore, Pesaro
  - AUSL Romagna - Ospedale Santa Maria dell Croci, Ravenna
  - Arcispedale Di S. Maria Nuova, Reggio Emilia
  - AUSL Romagna - Ospedale Infermi di Rimini, Rimini
  - H. San Giovanni - Addolorata, Roma
  - Universita Degli Studi Di Roma La Sapienza - Ospedale Sant'Andrea, Roma
  - Azienda Ospedallera Universitaria - Policlinico Tor Vergata, Rome
  - Instituto Regina Elena / Instituti Fisioterapici Ospitalieri, Rome
  - Ospedale San Eugenio, Rome
  - Clinica Ematologica dell'Universita di Roma La Sapienza, Rome
  - Ospedale Casa Sollievo Della Sofferenza, San Giovanni Rotondo
  - Azienda Ospedaliera Città della Salute e della Scienza di Torino - Ospedale Molinette, Torino
  - Azienda Ospedaliero-Universitaria "Santa Maria della Misericordia" di Udine, Udine
- Vilnius University Hospital Santariskiu Clinics, Vilnius, Lithuania
- Netherlands (8):
  - Rijnstate Hospital, Arnhem
  - Reinier De Graaf Gasthuis, Delft
  - Unversity Medical Center Groningen, Groningen
  - Medisch Centrum Leeuwarden-Zuid, Leeuwarden
  - Academisch Ziekenhuis Maastricht, Maastricht
  - Radboud University Medical Center Nijmegen, Nijmegen
  - Canisius-Wilhelmina Ziekenhuis, Nijmegen
  - HagaZiekenhuis - locatie Leyweg, The Hague
- Hospital Escolar Soa Joao, Porto, Portugal

REFERENCES:
- [Derived] Efficace F, Kicinski M, Coens C, Suciu S, van der Velden WJFM, Noppeney R, Chantepie S, Griskevicius L, Neubauer A, Audisio E, Luppi M, Fuhrmann S, Foa R, Crysandt M, Gaidano G, Vrhovac R, Venditti A, Posthuma EFM, Candoni A, Baron F, Legrand O, Mengarelli A, Fazi P, Vignetti M, Giraut A, Wijermans PW, Huls G, Lubbert M. Decitabine in older patients with AML: quality of life results of the EORTC-GIMEMA-GMDS-SG randomized phase 3 trial. Blood. 2024 Aug 1;144(5):541-551. doi: 10.1182/blood.2023023625. PMID 38717861
- [Derived] Lubbert M, Wijermans PW, Kicinski M, Chantepie S, Van der Velden WJFM, Noppeney R, Griskevicius L, Neubauer A, Crysandt M, Vrhovac R, Luppi M, Fuhrmann S, Audisio E, Candoni A, Legrand O, Foa R, Gaidano G, van Lammeren-Venema D, Posthuma EFM, Hoogendoorn M, Giraut A, Stevens-Kroef M, Jansen JH, de Graaf AO, Efficace F, Ammatuna E, Vilque JP, Wasch R, Becker H, Blijlevens N, Duhrsen U, Baron F, Suciu S, Amadori S, Venditti A, Huls G; EORTC Leukemia Group, GIMEMA, and German MDS Study Group. 10-day decitabine versus 3 + 7 chemotherapy followed by allografting in older patients with acute myeloid leukaemia: an open-label, randomised, controlled, phase 3 trial. Lancet Haematol. 2023 Nov;10(11):e879-e889. doi: 10.1016/S2352-3026(23)00273-9. PMID 37914482